CLINICAL TRIAL: NCT04370119
Title: Screening for SARS-CoV-2-Infections and Monitoring of Serological Responses to SARS-CoV-2 in Healthcare Workers
Brief Title: Screening for COVID-19 and Monitoring of Serological Responses to SARS-CoV-2 in Healthcare Workers
Acronym: SeCo
Status: Completed | Type: Observational
Sponsor: University Medicine Greifswald (Other)
Collaborators: Friedrich Loefler Institute for Animal Health (Unknown); EUROIMMUN AG (Unknown)
Responsible Party: Sponsor
Other Study IDs: BB 068/20
Record Dates: First submitted 2020-04-29; First posted 2020-04-30 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: SARS-CoV-2
Keywords: Serology; antibody formation; epidemiology; immunity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, nasal/throat swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- (1) Healthcare workers: All healthcare workers at University Medicine Greifswald who were enrolled in the study between 04/2020-08/2020
  Interventions: Diagnostic Test: Nasal swab; Diagnostic Test: Serum testing
- (2) Healthcare workers in high-risk areas of the hospital (intensive care, emergency medicine): Healthcare workers at University Medicine Greifswald who were enrolled in the study between 01/2021-03/2021
  Interventions: Diagnostic Test: Nasal swab; Diagnostic Test: Serum testing
- (3) Healthcare workers after SARS-CoV-2 vaccination: Healthcare workers at University Medicine Greifswald who received a SARS-CoV-2 vaccination within the last 7-21 days
  Interventions: Diagnostic Test: Nasal swab; Diagnostic Test: Serum testing

INTERVENTIONS:
Diagnostic Test: Nasal swab — SARS-CoV-2 PCR
Diagnostic Test: Serum testing — Anti-SARS-CoV2 S protein IgG ELISA, serological changes after SARS-CoV-2 vaccination

SUMMARY:
The main objectives of this study are 1) to establish the prevalence of SARS-CoV-2 in asymptomatic healthcare workers (HCWs) in an early phase of community spread as well as 2) to monitor the future spread of the disease by assessing serological responses to SARS-CoV-2 in symptomatic and asymptomatic HCWs over time and 3) to improve the assessment of the immune response and its protective effect as well as the assessment of infectivity of affected HCWs and 4) to evaluate the value and significance of antibody formation and serological antibody tests and 5) to be able to evaluate possible future preventive and / or therapeutic approaches against SARS-CoV-2, e.g. to assess vaccination effects

DETAILED DESCRIPTION:
This study aims to collect information on staff working at the Greifswald University hospital.

Over a 5 year period, a maximum of 12 study visits per participant are planned. At each visit, nasal/throat swabs (for PCR testing) and/or blood samples (to assess immunological responses, e.g. for SARS-CoV-2 antibody testing) will be collected. This will help to gain a better understanding of viral load and immunological responses, e.g. antibody development and their effects over time.

At study visit 2 - 12, participants will also be asked to fill in a questionnaire (asking for SARS-CoV-2 risk factors, perceived risk, impact of the pandemic on their quality of life, their interest in getting a SARS-CoV-2 vaccine/their SARS-CoV-2 vaccination status and vaccination side effects).

The remaining blood samples will be stored in a repository for future research.

The study is part of a modular SARS-CoV-2-research programme of the University Medicine Greifswald.

ELIGIBILITY:
Inclusion Criteria:

1. >= 18 years of age
2. Willing and able to complete a written consent form
3. Willing to have blood samples stored for future research
4. Healthcare worker employed at Greifswald University Hospital

Exclusion Criteria:

1. < 18 years of age
2. Decline to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Health Care Worker
Sampling Method: Non-Probability Sample
Enrollment: 1092 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2021-04-23 (Actual); Study Completion 2025-04-27 (Actual)

PRIMARY OUTCOMES:
Number of people with detectable antibodies to SARS-CoV-2 | 1 year
  Anti-SARS-CoV-2 S protein IgG ELISA/ Anti-SARS-CoV-2 NCP IgG ELISA

SECONDARY OUTCOMES:
Number of people with detectable SARS-CoV-2 nucleic acid | First study visit (baseline)
  SARS-CoV-2 PCR

OTHER OUTCOMES:
Number of people with detectable antibodies to SARS-CoV-2 | First study visit (baseline)
  Anti-SARS-CoV-2 S protein IgG ELISA/ Anti-SARS-CoV-2 NCP IgG ELISA
Number of people with detectable antibodies to SARS-CoV-2 | 2 years
  Anti-SARS-CoV-2 S protein IgG ELISA/ Anti-SARS-CoV-2 NCP IgG ELISA
Number of people with detectable antibodies to SARS-CoV-2 | 3 years
  Anti-SARS-CoV-2 S protein IgG ELISA/ Anti-SARS-CoV-2 NCP IgG ELISA
Number of people with detectable antibodies to SARS-CoV-2 | 4 years
  Anti-SARS-CoV-2 S protein IgG ELISA/ Anti-SARS-CoV-2 NCP IgG ELISA
Number of people with detectable antibodies to SARS-CoV-2 | 5 years
  Anti-SARS-CoV-2 S protein IgG ELISA/ Anti-SARS-CoV-2 NCP IgG ELISA
Number of people with detectable SARS-CoV-2 nucleic acid | 2 years
  SARS-CoV-2 PCR
Number of people with detectable SARS-CoV-2 nucleic acid | 3 years
  SARS-CoV-2 PCR
Number of people with detectable SARS-CoV-2 nucleic acid | 4 years
  SARS-CoV-2 PCR
Number of people with detectable SARS-CoV-2 nucleic acid | 5 years
  SARS-CoV-2 PCR
SARS-CoV-2 risk factors, perceived risk of infection, impact of the pandemic on quality of life, vaccination interest/vaccination status, vaccination side effects | 1 year
  As assessed by a questionnaire
SARS-CoV-2 risk factors, perceived risk of infection, impact of the pandemic on quality of life, vaccination interest/vaccination status, vaccination side effects | 2 years
  As assessed by a questionnaire
SARS-CoV-2 risk factors, perceived risk of infection, impact of the pandemic on quality of life, vaccination interest/vaccination status, vaccination side effects | 3 years
  As assessed by a questionnaire
SARS-CoV-2 risk factors, perceived risk of infection, impact of the pandemic on quality of life, vaccination interest/vaccination status, vaccination side effects | 4 years
  As assessed by a questionnaire
SARS-CoV-2 risk factors, perceived risk of infection, impact of the pandemic on quality of life, vaccination interest/vaccination status, vaccination side effects | 5 years
  As assessed by a questionnaire
Serological changes after SARS-CoV-2 vaccination | 7 days to 6 months after vaccination
  Serological changes after SARS-CoV-2 vaccination, cohort 3 only

CONTACTS AND LOCATIONS:
Overall Officials: Nils-Olaf Hübner, Prof.Dr., Principal Investigator — University Medicine Greifswald; Karsten Becker, Prof.Dr., Principal Investigator — University Medicine Greifswald
Locations (1):
- Greifswald University Medicine, Greifswald, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Esefeld M, Handtke S, Kaiser R, Nicolai L, Di Fina L, Rossaro D, Wesche J, Rath J, Wienrich AC, Hoffmann T, Harasser L, Feistritzer C, Loacker L, Lotfi K, Holmstrom M, Antovic J, Steil L, Volker U, Ulm L, Becker K, Hubner NO, Greinacher A, Thiele T. Platelet-activating histone/antihistone IgG complexes in anti-PF4-negative thrombosis and thrombocytopenia syndrome. Blood Adv. 2025 Aug 26;9(16):4323-4335. doi: 10.1182/bloodadvances.2024015076. PMID 40179418
- [Derived] Handtke S, Wolff M, Zaninetti C, Wesche J, Schonborn L, Aurich K, Ulm L, Hubner NO, Becker K, Thiele T, Greinacher A. A flow cytometric assay to detect platelet-activating antibodies in VITT after ChAdOx1 nCov-19 vaccination. Blood. 2021 Jul 1;137(26):3656-3659. doi: 10.1182/blood.2021012064. PMID 33945605